CLINICAL TRIAL: NCT04480944
Title: Massive Burns: Retrospective Analysis of Change in Outcomes Across 18 Years
Brief Title: Massive Burns: Retrospective Analysis of Changes in Outcomes Across 18 Years
Acronym: MassiveBurns
Status: Completed | Type: Observational
Sponsor: Mette M Berger (Other)
Responsible Party: Sponsor-Investigator, Mette M Berger, Associate professor, MD, PhD, Centre Hospitalier Universitaire Vaudois
Organization: Centre Hospitalier Universitaire Vaudois (Other)
Other Study IDs: CER2018-02268
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Burns
Keywords: Massive burns; Intensive care unit; Burn surgery; Burn infections; Skin grafts; Critical illness; Cultured epithelial autografts; Nutrition; Glucose
MeSH Terms: conditions — Burns; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Burns treatment and management has evolved since the 90s, particularly for massive burns (≥ 50% of total body surface area (TBSA)). This study aims at analyzing the impact of the management changes on the length of intensive care unit (ICU) stay, the take of skin grafts and the mortality.

DETAILED DESCRIPTION:
Review of all massively burned patients treated at Lausanne University Hospital burn intensive care unit (ca. 40-60 patients). Analysis of changes in length of intensive care unit stay (LICU), skin graft take rate or mortality between 2000 and 2018.

Hypothesis : the optimization of resuscitation procedures and of nutrition therapy combined with the use of novel surgical techniques has brought a significant improvement in outcomes.

Association between outcomes and year of admission will be assessed through correlation analysis and logistic regression analysis. Potential cofounders will be assessed through stepwise linear regression analysis

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (>18 years old) with burns ≥50% TBSA admitted in the burn intensive care unit (ICU) of the Lausanne University Hospital

Exclusion Criteria:

* Patients admitted in the burn center ICU with another primary diagnosis than burn (e.g. necrotizing fasciitis, gangrene, toxic epidermal necrolysis)
* Patients referred from and/or to another ICU
* Patients in which active withdrawal of care was decided within 48h of admission
* Patients with first degree burns only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients with extremely large burns (massive burn >50% TBSA) admitted and treated from beginning to end in the burn intensive care unit of a university hospital burn center in Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
LICU/Percent TBSA | 18 years
  Ratio between the length of stay in the ICU and the total body surface area burned

SECONDARY OUTCOMES:
Percent TBSA grafted/ Percent TBSA deep burns | 18 years
  Ratio between the TBSA grafted and the deep burns TBSA
Daily nutritional intakes | 18 years
  Daily energy, proteins, lipids and carbohydrates intakes per kilogram of body weight
Mortality | 18 years
  Percentage of patients who received maximal care and died nonetheless

CONTACTS AND LOCATIONS:
Overall Officials: Wassim Raffoul, MD, Study Director — CHUV
Locations (1):
- Adult ICU and Burn ICU, Lausanne University Hospital, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pantet O, Stoecklin P, Vernay A, Berger MM. Impact of decreasing energy intakes in major burn patients: A 15-year retrospective cohort study. Clin Nutr. 2017 Jun;36(3):818-824. doi: 10.1016/j.clnu.2016.05.007. Epub 2016 May 24. PMID 27256559
- [Background] Brusselaers N, Hoste EA, Monstrey S, Colpaert KE, De Waele JJ, Vandewoude KH, Blot SI. Outcome and changes over time in survival following severe burns from 1985 to 2004. Intensive Care Med. 2005 Dec;31(12):1648-53. doi: 10.1007/s00134-005-2819-6. Epub 2005 Oct 12. PMID 16220315